CLINICAL TRIAL: NCT04366791
Title: The RESCUE 1-19 Trial: Radiation Eliminates Storming Cytokines and Unchecked Edema as a 1-Day Treatment for COVID-19
Brief Title: Radiation Eliminates Storming Cytokines and Unchecked Edema as a 1-Day Treatment for COVID-19
Acronym: RESCUE 1-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI does not plan on putting any new patients on study. All patients completed this trial.
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mohammad K. Khan, Study Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000476; NCI-2020-02676 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD5002-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pneumonia; Coronavirus Infection in 2019 (COVID-19); Severe Acute Respiratory Syndrome (SARS) Pneumonia
MeSH Terms: conditions — Pneumonia; COVID-19; Severe Acute Respiratory Syndrome | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive care (low-dose radiation therapy) (Experimental): Patients undergo 1 fraction of low-dose radiation therapy.
  Interventions: Radiation: Low Dose Radiation Therapy

INTERVENTIONS:
Radiation: Low Dose Radiation Therapy — Undergo low-dose radiation therapy
  Other Names: Low Dose Radiation

SUMMARY:
This phase I/II trial studies low-dose radiation therapy as a focal anti-inflammatory treatment for patients with pneumonia or SARS associated with COVID-19 infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare treatment of COVID-19 between best supportive care plus provider's treatment choice versus best supportive care plus low-dose, whole-lung radiation therapy

OUTLINE:

Patients undergo 1 fraction of low-dose radiation therapy.

After completion of study treatment, patients are followed up at days 1-7, and 14 after last dose of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have had a positive test confirming the diagnosis of COVID-19
* Have had clinical signs of severe acute respiratory syndrome or pneumonia (dyspnea, cough, with need for oxygen support at the time of enrollment)
* Have visible consolidations/ground glass opacities on chest x-ray or computed tomography
* Have received pre-intubation respiratory support or undergone endotracheal intubation and have been on ventilator support for no longer than 5 (five) calendar days prior to the schedule date of delivery of low-dose radiation therapy.
* Willingness and ability of the subject to comply with scheduled visits, protocol-specified laboratory tests, other study procedures, and study restrictions
* Evidence of a signed informed consent/assent indicating that the subject is aware of the infectious nature of the disease and has been informed of the procedures to be followed, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* No use of disallowed medications 1 day prior to delivery of LDRT: Azithromycin, chloroquine, hydrochloroquine, COVID-targeted antiviral medications
* Pregnant and/or planned to be pregnant within in next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Rate of extubation (for intubated patients) | Screening up to 28 days after radiation therapy
  The rate will be reported, along with a two-sided 95% exact binomial confidence interval, using the Clopper-Pearson method. The observed extubation rate will be compared to the null rate of 20% using a two-sided binomial test. Statistical significance is assessed at the 0.05 level.

SECONDARY OUTCOMES:
Clinical outcome - Temperature | Screening up to 28 days after radiation therapy
  Temperature in degrees (F)
Clinical outcome - Heart Rate | Screening up to 28 days after radiation therapy
  Heart rate in beats per minutes
Clinical outcome - Systolic blood pressure | Screening up to 28 days after radiation therapy
  Systolic blood pressure in mm Hg
Clinical outcome - Oxygenation | Screening up to 28 days after radiation therapy
  Oxygen saturation in percentage
Clinical outcome - Respirations | Screening up to 28 days after radiation therapy
  Respiratory rate in breaths per minute
Clinical outcome - FiO2 | Screening up to 28 days after radiation therapy
  FI02 in percentage
Clinical outcome - PEEP | Screening up to 28 days after radiation therapy
  Positive end expiratory pressure (PEEP) in cm H20
Clinical outcome - Tidal volume | Screening up to 28 days after radiation therapy
  Tidal volume in mL
Clinical outcome - Intubation/Extubation events | Screening up to 28 days after radiation therapy
  Extubation/intubation events in percentage
Clinical outcome - Overall survival | Screening up to 28 days after radiation therapy
  Survival in percentage
Radiographic outcome - Chest xray | Screening up to 28 days after radiation therapy
  Serial chest x-rays categorized using published scale into ordinal ranks 1-5 for SARS.
Radiographic outcome - CT can | Screening up to 28 days after radiation therapy
  CT scans with volume of consolidation measured in cubic centimeters.
Serologic outcome - WBC | Screening up to 28 days after radiation therapy
  White blood cell count in cell count x 10^3/mcL
Serologic outcome - Hgb | Screening up to 28 days after radiation therapy
  Hemoglobin in gm/dL
Serologic outcome - Procalcitonin | Screening up to 28 days after radiation therapy
  Procalcitonin in ng/mL
Serologic outcome - ANC | Screening up to 28 days after radiation therapy
  Absolute neutrophil count in cell count x 10^3/mcL
Serologic outcome - Creatine kinase | Screening up to 28 days after radiation therapy
  Creatine kinase in units/L
Serologic outcome - Myoglobin | Screening up to 28 days after radiation therapy
  Myoglobin in ng/mL
Serologic outcome - Albumin | Screening up to 28 days after radiation therapy
  Albumin in gm/dL
Serologic outcome - PT/PTT | Screening up to 28 days after radiation therapy
  Coagulation pathway time in seconds
Serologic outcome - D-Dimer | Screening up to 28 days after radiation therapy
  D-Dimer in ng/mL
Serologic outcome - GGT | Screening up to 28 days after radiation therapy
  Gamma-glutamyl transferase in units/L
Serologic outcome -Triglycerides | Screening up to 28 days after radiation therapy
  Trygliciericdes in mg/dL
Serologic outcome -Ferritin | Screening up to 28 days after radiation therapy
  Ferritin in ng/mL
Serologic outcome -Fibrinogen | Screening up to 28 days after radiation therapy
  Fibrinogen in mg/dL
Serologic Immune markers flow cytometry | Screening up to 28 days after radiation therapy
  Immune marker flow cytometry (refractive index)
Serologic outcome -Bilirubin | Screening up to 28 days after radiation therapy
  Bilirubin in mg/dL
Serologic outcome - LDH | Screening up to 28 days after radiation therapy
  Lactate Dehydrogenase in units/L
Serologic outcome - Creatinine | Screening up to 28 days after radiation therapy
  Creatinine in mg/dL
Serologic outcome - EGFR | Screening up to 28 days after radiation therapy
  Estimated Glomerular Filtration Rate in mL/min/m2
Serologic outcome - CRP | Screening up to 28 days after radiation therapy
  C-Reactive Protein in mg/L
Serologic outcome - ALT | Screening up to 28 days after radiation therapy
  Alanine Aminotransferase in units/L
Serologic outcome - AST | Screening up to 28 days after radiation therapy
  Asparatate Aminotransferase in units/L
Serologic outcome - Troponin-I | Screening up to 28 days after radiation therapy
  Troponin-I in ng/mL
Serologic outcome - BNP | Screening up to 28 days after radiation therapy
  B-Natriuretic Peptid in pg/mL
Serologic outcome - Blood Gases pH | Screening up to 28 days after radiation therapy
  pH (no unit)
Serologic outcome - Blood Gases pO2 | Screening up to 28 days after radiation therapy
  pressure of O2 in mm Hg
Serologic outcome - Blood Gases pCO2 | Screening up to 28 days after radiation therapy
  pressure of CO2 in mm Hg
Serologic outcome - Lactic Acid | Screening up to 28 days after radiation therapy
  Lactic Acid in mmol/L
Serologic outcome - IL-6 | Screening up to 28 days after radiation therapy
  Interleukin-6 in pg/mL
Serologic outcome - Potassium | Screening up to 28 days after radiation therapy
  Potassium in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Khan, MD, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hosptial, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
No
  Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.

REFERENCES:
- [Derived] Hess CB, Eng TY, Nasti TH, Dhere VR, Kleber TJ, Switchenko JM, Weinberg BD, Rouphael N, Tian S, Rudra S, Taverna LS, Daisson AP, Ahmed R, Khan MK. Whole-lung low-dose radiation therapy (LD-RT) for non-intubated oxygen-dependent patients with COVID-19-related pneumonia receiving dexamethasone and/or remdesevir. Radiother Oncol. 2021 Dec;165:20-31. doi: 10.1016/j.radonc.2021.10.003. Epub 2021 Oct 13. PMID 34653525

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT04366791/Prot_SAP_000.pdf